CLINICAL TRIAL: NCT05757947
Title: Multicenter Clinical Trial of Myocardial Revascularization Using I-conduit and No-touch Saphenous Vein Graft
Brief Title: Study of the No-touch Saphenous Vein Graft
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Dmitry Khvan, candidate of medical sciences, senior researcher, сardiovascular surgeon of the NMRC named after academician E.N. Meshalkin of the Ministry of Health of Russian Federation, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Super-SVG
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis; Graft Failure; Cardiac Ischemia; Surgery
Keywords: no-touch saphenous vein graft; CABG
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "no-touch" saphenous vein as I-graft (Active Comparator): Coronary bypass surgery according to the I-graft method. Proximal anastomosis to RIMA.
  Interventions: Procedure: Сoronary bypass surgery according to the I-graft method
- "no-touch" saphenous vein as conventional free graft (Active Comparator): Coronary artery bypass grafting using the free conduit technique. Proximal anastomosis to aorta.
  Interventions: Procedure: Сoronary bypass surgery by the method of free conduit

INTERVENTIONS:
Procedure: Сoronary bypass surgery according to the I-graft method — Revascularization of the right coronary artery basin will be performed using "no-touch" SVG and the formation of an anastomosis of the stump of the right internal mammary artery and end-to-end saphenous vein graft.
  Arms: "no-touch" saphenous vein as I-graft
Procedure: Сoronary bypass surgery by the method of free conduit — Revascularization of the right coronary artery basin will be performed using "no-touch" SVG and anastomosis of the saphenous vein graft to aorta.
  Arms: "no-touch" saphenous vein as conventional free graft

SUMMARY:
Authors hypothesize that "no-touch" saphenous vein as I graft is superior over conventional "no-touch" saphenous vein as free graft in the incidence of graft patency.

DETAILED DESCRIPTION:
A multicenter single blind prospective randomized superiority study is conducted. Our hypothesis is that there is difference in the incidence of "no-touch" saphenous vein graft patency using it as the conventional free graft (group C) and I graft (group I) for myocardial revascularization more than 28%. If there is truly difference between groups, then total 106 patients for both groups are required to be 90% sure that the upper limit of a one-sided 95% confidence interval would reveal a difference in favour of the "no-touch" saphenous vein I graft of 28%. The blinding process is applied to a patient, who is informed about received harvesting method of saphenous vein, but don't know the type of the graft cofiguration. The study was approved by Institutional Review Board. Depending on a type of the procedure, the patients are divided into two groups: conventional free graft (group C) 53 patients and I graft (group I) 53 patients. Randomization is conducted befor operation by using accidental sampling.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease requiring three-vessel myocardial revascularization
* Patient consent to the study

Exclusion Criteria:

* The diameter of the target arteries for conduits of the internal mammary arteries is less than 1 mm
* Hemodynamically significant atherosclerosis of the subclavian arteries in the first segment
* Stenosis of the right coronary artery less than 90%
* Concomitant pathology requiring additional simultaneous surgical correction
* Lack of IMA
* COPD with FEV1 <60%
* BMI >35
* Prior heart surgery
* Oncological diseases with a life expectancy of less than 5 years
* ACS
* CKD stage 4 and higher
* The diameter of the SVG is less than 2 mm or its varicose expansion is more than 6 mm
* CLTI IIb and more
* Atherosclerosis of the brachiocephalic artery more than 50%

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Patency of "no-touch" saphenous vein graft | 12 months after surgery
  Assessment of the patency of coronary shunts

SECONDARY OUTCOMES:
Recurrence of angina pectoris | 6 and 12 months after after surgery
  Estimated percentage of participants with symptomatic angina at 6 and 12 months after surgery
MACE | 6 and 12 months after after surgery
  Estimated percentage of participants with major adverse cardiac events at 6 and 12 months post-surgery
Complications of the conduit fence site | 6 and 12 months after after surgery
  Estimated percentage of participants with wound complications, development of wound infection, postoperative neurological complications at the sampling site at 6 and 12 months after surgery
Survival rate | 6 and 12 months after after surgery
  Estimated percentage of participants who died at 6 and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Khvan, Ph.D., Principal Investigator — NMCR named after academician E.N. Meshalkin of the Ministry of Health of rhe Russian
Locations (1):
- NMCR named after academician E.N. Meshalkin of the Ministry of Health of rhe Russian, Novosibirsk, Novosibirsk Oblast, Russia